CLINICAL TRIAL: NCT00855127
Title: Early Biomarkers of Acute Kidney Injury in Liver Transplant Patients
Brief Title: New Urine and Blood Markers for Acute Kidney Injury in Liver Transplant Patients
Status: Withdrawn | Type: Observational
Why Stopped: no enrollment
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Washington (Other); Denver Health Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0769
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Renal Insufficiency, Acute
Keywords: Biological Markers; Renal Replacement Therapy; Mortality
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine supernatent Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplant recipients

SUMMARY:
The purpose of this study is to find new blood and urine tests that detect acute kidney injury earlier than our current blood tests in patients receiving a liver transplant.

DETAILED DESCRIPTION:
Patients with end stage liver disease that receive a liver transplant will be studied to determine if novel serum and urine biomarkers (serum cystatin C, urine interleukin-18 [IL-18] and urine neutrophil gelatinase associated lipocalin [NGAL]) can predict the outcome measures listed above.

ELIGIBILITY:
Inclusion Criteria:

* First time liver transplant recipient
* Cadaveric or living donor livers

Exclusion Criteria:

* Unconscious patients or patients who cannot give consent
* Pregnant women
* Prisoners
* Patients receiving dialysis before or during liver transplant operation
* Patients receiving simultaneous liver-kidney transplants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the University of Colorado Hospital or the University of Washington Medical Center for a liver transplant operation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Development of acute kidney injury as defined by a 50% increase in serum creatinine | Within 2 to 5 days of liver transplant that is sustained for at least 24 hours

SECONDARY OUTCOMES:
Development of severe acute kidney injury, as defined as a doubling of serum creatinine | Within 2-5 days of transplant that is sustained for at least 24 hours
The need for renal replacement therapy | After liver transplant operation to discharge
All cause mortality | After liver transplant operation to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Walcher, MD, Principal Investigator — University of Colorado, Denver; Charles L Edelstein, MD, PhD, Study Director — University of Colorado, Denver; Connie L Davis, MD, Study Director — University of Washington
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Edelstein CL. Biomarkers of acute kidney injury. Adv Chronic Kidney Dis. 2008 Jul;15(3):222-34. doi: 10.1053/j.ackd.2008.04.003. PMID 18565474
- [Background] Parikh CR, Mishra J, Thiessen-Philbrook H, Dursun B, Ma Q, Kelly C, Dent C, Devarajan P, Edelstein CL. Urinary IL-18 is an early predictive biomarker of acute kidney injury after cardiac surgery. Kidney Int. 2006 Jul;70(1):199-203. doi: 10.1038/sj.ki.5001527. Epub 2006 May 17. PMID 16710348
- [Background] Parikh CR, Abraham E, Ancukiewicz M, Edelstein CL. Urine IL-18 is an early diagnostic marker for acute kidney injury and predicts mortality in the intensive care unit. J Am Soc Nephrol. 2005 Oct;16(10):3046-52. doi: 10.1681/ASN.2005030236. Epub 2005 Sep 7. PMID 16148039